CLINICAL TRIAL: NCT01171469
Title: Phase I Study of Vaccination With Dendritic Cells Loaded With Brain Tumor Stem Cells for Recurrent or Progressive Malignant Gliomas
Brief Title: Vaccination With Dendritic Cells Loaded With Brain Tumor Stem Cells for Progressive Malignant Brain Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008LS053; 0809M48641 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Brain Tumor; Glioblastoma; Medulloblastoma; Ependymoma; Anaplastic Astrocytoma
Keywords: Brain tumor; Immunotherapy; Glioma
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma; Medulloblastoma; Ependymoma; Astrocytoma; Glioma | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dose Level 3 (Experimental): 15 Million dendritic cells (DCs) - administered via intradermal injections in 0.5 ml Phosphate Buffered Saline (PBS) in the shoulders near the back of the neck to facilitate trafficking of the DCs to the cervical lymph nodes.
  Interventions: Biological: Dendritic Cells; Drug: Imiquimod
- Dose Level 2 (Experimental): 10 Million dendritic cells (DCs) - administered via intradermal injections in 0.5 ml Phosphate Buffered Saline (PBS) in the shoulders near the back of the neck to facilitate trafficking of the DCs to the cervical lymph nodes.
  Interventions: Biological: Dendritic Cells; Drug: Imiquimod
- Dose Level 1 (Experimental): 5 Million dendritic cells (DCs) - administered via intradermal injections in 0.5 ml Phosphate Buffered Saline (PBS) in the shoulders near the back of the neck to facilitate trafficking of the DCs to the cervical lymph nodes.
  Interventions: Biological: Dendritic Cells; Drug: Imiquimod

INTERVENTIONS:
Biological: Dendritic Cells — 5, 10 or 15 Million dendritic cells (DCs) - administered via intradermal injections in 0.5 ml Phosphate Buffered Saline (PBS) in the shoulders near the back of the neck to facilitate trafficking of the DCs to the cervical lymph nodes.
  Other Names: DCs
Drug: Imiquimod — Imiquimod (INN) is a prescription medication that acts as an immune response modifier. Imiquimod is marketed as 5% Aldara cream in 250 mg packets, providing a total dose of 12.5 mg per packet and sufficient to cover 20 square centimeters. The contents of ½ of a packet will be applied as a thin film to cover approximately 10 square centimeters of skin in the area of the planned vaccination.
  Other Names: Aldara

SUMMARY:
This is a single center Phase I study to determine the safety and maximum tolerated dose (MTD) of autologous dendritic cells (DCs) loaded with allogeneic brain tumor stem cells administered as a vaccination in children and adults with recurrent brain tumors. Once the MTD has been determined, we will conduct a phase II study to determine efficacy.

Clinical trials that utilize DCs for immunotherapy have demonstrated significant survival benefit for patients who exhibit robust immune responses against tumor cells. Unfortunately, at the present time the majority of tumor patients are unable to mount an adequate immune response and thus succumb to their tumors. We postulate that the inability to generate an appropriate immune response in these patients is due to a lack of sufficient numbers of appropriate T cells due to an inadequate source of tumor antigens.

DETAILED DESCRIPTION:
Autologous DCs will be obtained from peripheral blood mononuclear cells (PBMCs) from each patient by leukapheresis. An established BTSC line will be used as an allogeneic source of tumor antigen. Approximately 4 weeks will be required after the leukapheresis for vaccine production and the first vaccine administration.

Each patient will receive an injection of DCs at his/her assigned dose once every 2 weeks during the first 8 weeks, followed by injections every 4 weeks for an additional 10 vaccinations. Imiquimod will be applied to the vaccination site just prior to and 24 hours after each vaccine administration.

This study will use an accelerated dose escalation design (1 subject per level) until dose limiting toxicity (DLT) is encountered, after which a traditional phase I design (3 subjects per level) will be implemented. DLT is defined as grade 3 or greater treatment related toxicity. A total of 6 patients will be treated at the maximum tolerated dose (MTD) or, in the absence of DLT, at dose level 3.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed brain tumors (glioblastoma multiforme, anaplastic astrocytoma, medullo
* Age 0 through 17 years (pediatric subjects), and 18 years and above (adult subjects)
* Lansky score of ≥ 60 (0-15 years) or Karnofsky (16 years or older) performance score of ≥ 60%
* Adequate organ function within 14 days of study registration including the following:

  * Adequate bone marrow reserve: absolute neutrophil (segmented and bands) count (ANC) ≥ 1.0 x 10^9/L, platelets ≥100 x 10^9/L; hemoglobin ≥ 8 g/dL
  * Hepatic: bilirubin ≤1.3 mg/dL or 0-22 mmol/L, aspartate transaminase (AST) and alanine transaminase (ALT) < 3 x upper limit of normal (ULN)
  * Renal: Normal serum creatinine for age (below) or creatinine clearance >60 ml/min/1.73 m^2.
* Sexually active women of child bearing potential must agree to use adequate contraception (diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.) for the duration of the vaccination period. Sexually active men must agree to use barrier contraceptive for the duration of the vaccination period.
* Willingness to travel to participate in study if from outside local region.
* Voluntary written informed consent must be obtained from all patients (if of assent age) and their parents or legal guardians before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion criteria:

* Pregnant or breast-feeding. Pregnancy testing will be performed on all menstruating females within 14 days of study enrollment.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
* Currently receiving any other investigational agents.
* History of immune system abnormalities such as hyperimmunity (e.g., autoimmune diseases) and hypoimmunity (e.g., myelodysplastic disorders, marrow failures, AIDS, ongoing pregnancy, transplant immuno-suppression).
* Any conditions that could potentially alter immune function (e.g., AIDS, multiple sclerosis, diabetes, renal failure).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-09; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 4 Weeks Post Vaccination
  To determine the safety and maximum tolerated dose (MTD) of dendritic cells (DCs) loaded with brain tumor stem cells (BTSCs) as a source of tumor antigen for immunotherapy in children and adults with recurrent GBM, ependymoma or medulloblastoma brain tumors. Toxicity is determined using the criteria established by the National Cancer Institute's Common Terminology Criteria for Adverse Events V 4.0 (CTCAE).

SECONDARY OUTCOMES:
Time to Tumor Progression | Every 4 Weeks From Baseline to 1 Year
  To determine time to tumor progression in this patient population - exhibit a prolonged time to tumor progression by the absence of tumor growth as determined by MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Moertel, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States